CLINICAL TRIAL: NCT00600249
Title: Phase II Pilot Study Evaluating the Neoadjuvant Combination "Taxotere (Docetaxel) and Erbitux (Cetuximab) in Operable and "Triple Negative" Breast Cancer Patients. TENEO Study.
Brief Title: Assessment of the Efficacy of a Neoadjuvant Combination: "Chemotherapy-targeted Therapy" in Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TENEO
Record Dates: First submitted 2008-01-14; First posted 2008-01-24 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer.; Triple negative.; Neoadjuvant chemotherapy.; Targeted therapy.
MeSH Terms: conditions — Breast Neoplasms | interventions — Cetuximab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetuximab — dosage : 5mg/ml one administration per week: 400 mg/m2 then 250 mg/m2 during 18 weeks
  Other Names: Current sponsor code: EMD271786
Drug: Docetaxel — 100mg/m2 every 21 days 6 cycles of 21 days
  Other Names: CAS: 148408-66-6

SUMMARY:
The purpose of this study is to assess the pathological response rate in operable breast cancer patients treated by neoadjuvant combination "Taxotere-Erbitux".

ELIGIBILITY:
Inclusion Criteria:

* § Age > or equal to 18 years.§
* Performance status inferior or equal to 1 (WHO criteria)
* Histologically proven breast cancer, non metastatic, with clinical tumor diameter > or equal to 2 cm.
* HR negative and HER 2 negative.
* Clinical stage II and IIIa.
* Non prior treated patients either by surgery, radiotherapy, hormonotherapy or chemotherapy.§
* Adequate hematological, renal and hepatic functions : neutrophils > 2.109 /L, platelets > 100.109 /L, Hb > 10 g/dL, normal bilirubin, ASAT and ALAT inferior or equal to 2,5 ULN (upper normal limit), alkaline phosphatases £ 2,5 ULN, creatinine < 140 µmol/L or creatinine clearance > 60 mL/min.§
* Written informed consent§
* Affiliation with social security system (or profit being of such a mode) according to terms' of the law of August 9, 2004.

Exclusion Criteria:

* Male patient.
* Pregnant or lactating women or childbearing potential with no efficacy contraception.
* Other breast cancer form and particularly inflammatory form and/or negliged (T4b or T4d).§
* Non measurable tumor.
* Prior surgery or primary axillary dissection.
* Prior treatment for this new breast cancer.
* Under guardianship patient
* Patient with antecedent of second cancer, excepted in situ uterine carcinoma or baso-cellular cutaneous cancer considered as definitively cured.
* Patient with an associated pathology considered incompatible with the study.§ Cardiac, renal, medullar, respiratory or hepatic insufficiency.
* Significant neurological or psychiatric troubles.§ Symptomatic or evolutive troubles in CNS or metastasis.
* Peripheral neuropathy > grade 2 NCI-CTC (version 3.0)
* Previous allergy with polysorbate 80.
* Concomitant treatment with a drug tested in a clinical trial, participation to another clinical study, for the last thirty days or prior chemotherapy.
* Patients non stable for the following 6 months or leaving at a great distance of the participating center.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pathological complete response assessment of Taxotere-Erbitux combination | After 18 weeks of treatment

SECONDARY OUTCOMES:
Clinical, mammographic and ultrasound response Breast cancer conservation rate Overall and disease free survival Safety to treatments | After 18 weeks of treatment, at surgery and at five years (survival)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Chollet, MD, Principal Investigator — Centre Jean Perrin
Locations (6):
- France (6):
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU Albert Michallon, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier, Montluçon
  - Institut de Cancérologie de la LOIRE, Saint-Priest-en-Jarez
  - Hôpital Georges Pianta, Thonon-les-Bains

REFERENCES:
- [Derived] Nabholtz JM, Chalabi N, Radosevic-Robin N, Dauplat MM, Mouret-Reynier MA, Van Praagh I, Servent V, Jacquin JP, Benmammar KE, Kullab S, Bahadoor MR, Kwiatkowski F, Cayre A, Abrial C, Durando X, Bignon YJ, Chollet P, Penault-Llorca F. Multicentric neoadjuvant pilot Phase II study of cetuximab combined with docetaxel in operable triple negative breast cancer. Int J Cancer. 2016 May 1;138(9):2274-80. doi: 10.1002/ijc.29952. Epub 2015 Dec 28. PMID 26649807